CLINICAL TRIAL: NCT03855839
Title: The Effect of Posture Shirts on Posture During Functional Tasks in Healthy Participants.
Brief Title: The Effect of Posture Shirts on Posture During Functional Tasks
Status: Completed | Type: Observational
Sponsor: University College of Northern Denmark (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Other Study IDs: FOU-UU-2018-12_Sub-project1
Record Dates: First submitted 2019-02-13; First posted 2019-02-27 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: Posture; Muscle activity; Posture corrective shirts

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy participants: Participants will be ask to perform a repetitive upper limb task while posture is being monitored.This will be done while wearing a posture shirt, compression shirt or no shirt.
  Interventions: Device: Posture shirt; Device: Compression shirt

INTERVENTIONS:
Device: Posture shirt — Posture shirts are designed, and marketed to the general public and health service providers to improve posture and consequently alter muscle activity, reduce musculoskeletal pain and discomfort.
Device: Compression shirt — Compression shirts are designed for recreational sport activities and can be bought in any local sports store

SUMMARY:
This study investigates the effect of a posture shirt on posture during functional tasks such as office work.

DETAILED DESCRIPTION:
Poor posture have historically been blamed for pain and disability in the general population. A treatment-strategy that have gain popularity in recent years is the use of a posture shirt which is a compressive shirt designed and marketed to the general public and health service providers as a way to improve posture and consequently alter muscle activity, reduce musculoskeletal pain and discomfort. This study will investigate the effect of posture shirts on posture.

ELIGIBILITY:
Inclusion Criteria: - Healthy participants

* Pain free healthy participants
* Able to speak, read and understand Danish Exclusion Criteria: - Healthy participants
* Pain from the back, neck or shoulder area during the past 3 months
* Any discomfort in relation to computer use
* Lack of ability to cooperate

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male participants
Study Population: Healthy male participants
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-05-08 (Actual)

PRIMARY OUTCOMES:
Posture | Within session (2hr)
  Posture will be determined by measuring head and shoulder angles during a functional task

SECONDARY OUTCOMES:
Experienced pain | Within session (2hr)
  Any potential pain during the functional tasks will be monitored using a 0-11 numeric rating scale (NRS) with 0 being no pain and 10 being worst imaginable pain.
Concentration during task | Within session (2hr)
  Two questions regarding concentration during task was asked: (Q1: I had to concentrate to do the task, Q2: My concentration was constant throughout the task) were scores using a 5 point Likert scale (1: Strongly disagree; 2: Disagree; 3: Neither agree nor disagree; 4: Agree; 5: Strongly agree).
Consciousness of posture during task | Within session (2hr)
  Two questions regarding consciousness of posture during task was asked (Q1: I was conscious about how I was sitting in the beginning of the task , Q2: I was conscious about how I was sitting at the end of the task) was scored using a 5 point Likert scale (1: Strongly disagree; 2: Disagree; 3: Neither agree nor disagree; 4: Agree; 5: Strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Steffan W Christensen, PhD, Principal Investigator — Department of Physiotherapy, University College of Northern Denmark
Locations (1):
- Department of Physiotherapy, University College of Northern Denmark, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided